CLINICAL TRIAL: NCT01562015
Title: A Single Arm, Phase 2 Study of Ganetespib in Subjects With Advanced Non-Small-Cell Lung Cancer With Anaplastic Lymphoma Kinase Gene Rearrangement (ALK-Positive NSCLC)
Brief Title: A Study of Ganetespib in Subjects With ALK-Positive Non-Small-Cell Lung Cancer (NSCLC)
Acronym: CHIARA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-09
Record Dates: First submitted 2012-03-14; First posted 2012-03-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ganetespib (Experimental): Ganetespib IV infusion once per week for three consecutive weeks followed by a 1 week dose-free interval
  Interventions: Drug: Ganetespib

INTERVENTIONS:
Drug: Ganetespib — Ganetespib 200 mg/m2 administered 1 time per week for the first three weeks of a four week treatment cycle (Days 1, 8, and 15 of the 28 Day treatment cycle).

SUMMARY:
Phase 2 study of subjects with ALK positive, advanced NSCLC who have failed up to 3 prior therapies. The study will take place globally at multiple study centers. Subjects will be enrolled to receive ganetespib one time per week for three weeks followed by a rest week; and will repeat this schedule until the cancer gets worse or the subject is unable to tolerate ganetespib. The primary goal of the study is to determine how ganetespib is tolerated and how active it is in ALK positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older
* Pathological confirmation of advanced NSCLC
* Evidence of a translocation or an inversion event involving the ALK gene locus
* ECOG Performance Status 0 or 1

Exclusion Criteria:

* Prior therapy with ALK-targeted agents
* Prior treatment with Hsp90 inhibitor
* Known EGFR activating mutation
* Presence of active or untreated central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 1 year

SECONDARY OUTCOMES:
Duration of Response | 1 year
Disease Control Rate | 6 weeks and 12 weeks
Adverse events | 1 year
Progression Free Survival | From the date of study drug start until the date of first documented progression or date of death from any cause, whichever comes frist, assessed up to 3 years
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Synta Pharmaceuticals Investigative Site, Tampa, Florida
  - Synta Pharmaceuticals Investigative Site, Cleveland, Ohio
- Canada (3):
  - Synta Pharmaceuticals Investigative Site, Hamilton, Ontario
  - Synta Pharmaceuticals Investigative Site, Ottawa, Ontario
  - Synta Pharmaceuticals Investigative Site, Toronto, Ontario